CLINICAL TRIAL: NCT01735149
Title: Efficacy and Safety of Kochujang Pills on Improvement of Blood Lipids
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SRCM-HL-KOCHUJANG
Record Dates: First submitted 2012-11-23; First posted 2012-11-28 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kochujang Pills (Experimental)
  Interventions: Dietary Supplement: Kochujang Pills
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Kochujang Pills — Kochujang Pills (34.5g/day)
  Arms: Kochujang Pills
Dietary Supplement: Placebo — Placebo (34.5g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 12-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Kochujang pills on improvement of blood lipids. The investigators measured improvement of blood lipids parameters , including Total Cholesterol, LDL-C, Triglyceride and HDL-C, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-55 years old
* Total Cholesterol 200~260 mg/dl or LDL-C 110~190 mg/dl
* Able to give informed consent

Exclusion Criteria:

* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Total Cholesterol | 12 weeks
  Total cholesterol was measured in study visit 1(0 week) and visit 3(12 week).
Changes in LDL-C (LDL Low Density Lipoprotein-cholesterol) | 12 weeks
  LDL-C (LDL Low Density Lipoprotein-cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).

SECONDARY OUTCOMES:
Changes in Triglyceride | 12 weeks
  Triglyceride was measured in study visit 1(0 week) and visit 3(12 week).
Changes in HDL-C(High Density Lipoprotein-cholesterol) | 12 weeks
  HDL-C(High Density Lipoprotein-cholesterol) was measured in study visit 1(0 week) and visit 3(12 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea